CLINICAL TRIAL: NCT06542341
Title: Study to Evaluate the Efficacy of the décoLITE LED Device in Treating the Signs of Skin Aging of the décolletage Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Baker (Industry)
Responsible Party: Sponsor-Investigator, Steven Baker, Clinical trials Manager, Ismart
Organization: Ismart (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-5574 1/15/19
Record Dates: First submitted 2024-07-31; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Wrinkle

STUDY DESIGN:
Intervention Model Description: Open-label, single-centre trial.
Masking Description: Blinded photography- images masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active Light treatment Arm (Experimental): Treatment with red and near infra red light 5 x week for 6 weeks
  Interventions: Device: decoLITE (TN2037)

INTERVENTIONS:
Device: decoLITE (TN2037) — Red/Near infra red light therapy

SUMMARY:
To assess the efficacy of the décoLITE LED system in reducing the signs of skin aging of the décolletage area one week after a six-week treatment course.

DETAILED DESCRIPTION:
This was an open-label, single-center trial. Subjects carried out 5 treatments on separate days each week for 6 weeks. The plan for the study was to recruit 25 subjects to consider any dropouts to arrive at a final study total of 20.

Treatments were of 10 minutes duration using a combination of red (630nm) and near infrared (830nm) emitted from light emitting diodes. The device emitted 30mW/cm2 of light, delivering a dose of 18J/cm2 per treatment.

Subjects were assessed at baseline, at 5 weeks, and at 7 weeks (one week after the last treatment).

Assessments included separate evaluations of lines and pigment of the décolletage using the validated scale developed by Landau et al. by the principal investigator and a third party blinded physician, standardized photography, and recording of safety incidents. Subjective responses were based on treatment efficacy and ease of use of the device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female, 30 to 65 years of age.
* Fitzpatrick phototype I-VI skin.
* Gave written informed consent.
* Photoaging of the décolletage area.
* Agreed NOT to use anti-aging products that contain active ingredients such as retinol and glycolic acid on the treatment area during the study period.
* Agreed NOT to undergo any aesthetic treatments (such as chemical peels, microdermabrasion, laser surfacing, etc.) in the treatment area during the study period

Exclusion Criteria:

* Suffering from a systemic photosensitive disorder such as Lupus erythematosus, photosensitive eczema, or Albinism.
* Currently taking (or with a history of taking) medication that is known to induce photosensitivity.
* Having known malignancy and/or undergoing chemotherapy, radiotherapy, or high doses of corticosteroids.
* Suffering from keloid scars or birth marks in the treatment area.
* Suffering from eczema, psoriasis, or skin rashes in the treatment area.
* Had used an anti-aging product within the 4 weeks prior to commencing the study.
* Underwent plastic surgery within the last 6 months.
* Pregnant, breast-feeding, or wishing to become pregnant during the study period.
* Being enrolled in another clinical trial during the same study period.
* Having a planned hospital admission and/or surgical procedure for an illness or disease which existed before enrollment into the clinical trial, and which may interfere with the course or outcome of the study.
* Having medical or psychological condition(s) associated with a risk of poor protocol compliance (e.g., alcoholism or drug abuse).
* Undergoing or is likely to undergo other treatments of the décolletage area.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Reduction in chest lines at rest | 7 weeks after first treatment intervention
  Reduction in chest lines at rest according to the validated Merz aesthetics décolleté grading scale developed by Landau, et al (2016).

SECONDARY OUTCOMES:
Reduction in chest pigmentation | 7 weeks after first treatment intervention
  Reduction in chest pigmentation according to the validated Merz aesthetics décolleté grading scale developed by Landau, et al (2016

CONTACTS AND LOCATIONS:
Locations (1):
- Suite A, Astor House, Sutton Coldfield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share- confidential regulatory data